CLINICAL TRIAL: NCT06899633
Title: Multicenter, Observational, Descriptive Study of the Diagnosis, Course and Treatment of Patients With SLE in Routine Practice in Kazakhstan: a Registry Study With Retrospective and Prospective Components.
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00087
Record Dates: First submitted 2025-03-26; First posted 2025-03-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Description of SLE Activity in Patients in Routine Practice in the Republic of Kazakhstan; Description of the Course of SLE in Patients in the Republic of Kazakhstan; Description of Methods and Approaches to the Treatment of Patients With SLE in the Republic of Kazakhstan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Multicenter, observational, descriptive study of the diagnosis, course and treatment of patients with SLE in routine practice in Kazakhstan: a registry study with retrospective and prospective components.

DETAILED DESCRIPTION:
Primary Endpoints

1. Proportion of patients with varying SLE activity assessed by the SLEDAI 2K Activity Index at visits 0, 1, and 2
2. Proportion of patients with PGA changes in dynamics
3. Proportion of patients with changes in dynamics in general clinical tests from baseline data (Visit 0) at visits 1 and 2
4. Proportion of patients with varying SLE organ damage assessed by SLICC/ACR Damage Index - SLICC/ACR DI - SDI at visits 0, 1, and 2;
5. Proportion of patients with prescribed average daily dose of oral corticosteroids at visits 0, 1 and 2

   * Prednisone (and equivalents) = 0 mg/day
   * Patients with corticosteroids >0, but less than 5 mg/day; mean daily dose of oral corticosteroids
   * Patients with corticosteroids >5 mg/day: mean daily dose of oral corticosteroids
6. Proportion of patients treated with each line of treatment [13] at visits 0, 1, and 2

   * Glucocorticoids;
   * Cytostatics;
   * NSAIDs;
   * Biological drugs;
   * Immunoglobulins;
   * Other significant drugs that affect the course of treatment.

Secondary Endpoints :

1. Proportion of each sex among patients with SLE 2. Proportion of patients in different age groups 3. Proportion of patients of different races 4. Proportion of patients belonging to different nationalities 5. Proportion of patients with different social status groups 6. Proportion of patients in different BMI classes [9] 7. Proportion of patients with different ages of SLE onset and disease duration at diagnosis

* SLE course (relapsing-remitting, chronically active course; SLE remission)
* SLE disease activity (high, moderate, low)
* Average number of SLE exacerbations in the past year;
* Number and reasons for SLE-related hospitalizations and emergency department visits [11]
* Number and reasons for non-SLE-related hospitalizations;
* Number and percentage of patients with affected organs (kidneys, lungs, heart, nervous system, hematopoietic system, skin [10])
* Changes in the Revised Cutaneous Lupus Erythematosus Disease Areas and Severity Index (R-CLASI) scores 8 Dynamics of treatment results in patients with SLE:
* proportion of patients who achieved remission;
* proportion of patients with a decrease in the degree of SLE activity;
* proportion of patients who achieved low disease activity;
* proportion of patients with various reasons for stopping therapy
* proportion of patients switching drugs 9. Changes in quality of life indicators based on quality of life questionnaires and the presence of fatigue: Questionnaire (LupusQoL) for SLE at visits 0, 1 and 2.

  10. Proportion of patients achieving the combined endpoint LLDAS7.5 at baseline, visits 0, 1, and 2 (LLDAS with prednisone equivalent needed for response ≤ 7.5 mg/day) 11. Proportion of patients achieving the combined endpoint LLDAS5 at baseline, visits 0, 1, and 2 (LLDAS with prednisone equivalent needed for response ≤ 5 mg/day) 12. Proportion of patients achieving clinical remission at baseline, visits 0, 1, and 2.

  13. Changes in symptoms and clinical manifestations in patients with SLE 14. Changes in complications in patients with SLE 15. Proportion of patients with lupus nephritis 16. Changes in non-specific laboratory parameters (at visits 1 and 2 from the initial (visit 0)):
  * Complete blood count (CBC);
  * Complete urine count (CUA);
  * Coagulogram;
  * biochemical blood test: creatinine, total protein, ALT, AST, total bilirubin, total cholesterol, glucose;
  * CRP
  * GFR 17. Changes in immunological criteria:
* Indicators of C3, C4 components of the complement system at visits 0.1 and 2;
* IgG antibodies to double-stranded (native) DNA at visits 0, 1 and 2
* Antinuclear factor on the HEp-2 cell line (ANF) at visits 0 and 2 18. The proportion of patients adherent to treatment based on the Morisky-Green Questionnaire 19. The proportion of patients who had hospitalization and/or an emergency department visit [11] 20. The percentage of various reasons for SLE and non-SLE hospitalizations

ELIGIBILITY:
Inclusion Criteria

* Men and women aged 18 years and older with a verified diagnosis of SLE
* Patient signed and dated written informed consent form (ICF) by ICH GCP and local legislation prior to inclusion in the study for the prospective observational group.

Exclusion Criteria

* Absence of a signed consent form (ICF) in patients
* Cognitive impairments that hinder understanding the study objectives and completing questionnaires
* Participation in any randomized controlled clinical trial within 3 months prior to inclusion or during participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This non-interventional, multicenter observational study will enroll 500 adult patients with established SLE who are being followed and treated by rheumatologists in approximately 10 outpatient sites in approximately 8 regions of Kazakhstan.
  Eligible patients will be recruited sequentially during routine hospital visits. There will be no patient recruitment restrictions per site or region (to minimize selection bias at each site).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with varying SLE activity assessed by the SLEDAI 2K Activity Index at visits 0, 1, and 2 | 12 months
  Proportion of patients with varying SLE activity assessed by the SLEDAI 2K Activity Index at visits 0, 1, and 2
Proportion of patients with PGA changes in dynamics | 12 months
  Proportion of patients with PGA changes in dynamics
Proportion of patients with changes in dynamics in general clinical tests from baseline data (Visit 0) at visits 1 and 2 | 12 months
  Proportion of patients with changes in dynamics in general clinical tests from baseline data (Visit 0) at visits 1 and 2
Proportion of patients with varying SLE organ damage assessed by SLICC/ACR Damage Index - SLICC/ACR DI - SDI at visits 0, 1, and 2 | 12 months
  Proportion of patients with varying SLE organ damage assessed by SLICC/ACR Damage Index - SLICC/ACR DI - SDI at visits 0, 1, and 2
Proportion of patients (P) with prescribed average daily dose (dd) of oral corticosteroids(OC) at visits 0, 1 and 2 • Prednisone = 0 mg/day • P with OC >0 mg/day; mean dd of OC • P with OC >5 mg/day: mean dd of OC• P with OC ≤5 mg/day: mean dd of OC | 12 months
  Proportion of patients with prescribed average daily dose of oral corticosteroids at visits 0, 1 and 2
  * Prednisone (and equivalents) = 0 mg/day
  * Patients with corticosteroids >0 but less than 5 mg/day; mean daily dose of oral corticosteroids
  * Patients with corticosteroids >5 mg/day: mean daily dose of oral corticosteroids prescribed average daily dose (dd) of oral corticosteroids(OC) at visits 0, 1 and 2 • Prednisone = 0 mg/day • P with OC >0 mg/day; mean dd of OC • P with OC >5 mg/day: mean dd of OC• P with OC ≤5 mg/day: mean dd of OC
Proportion of patients treated with each line of treatment [13] at visits 0, 1, and 2 • Glucocorticoids; • Cytostatics; • NSAIDs; • Biological drugs; • Immunoglobulins; • Other significant drugs that affect the course of treatment | 12 months
  Proportion of patients treated with each line of treatment [13] at visits 0, 1, and 2
  * Glucocorticoids;
  * Cytostatics;
  * NSAIDs;
  * Biological drugs;
  * Immunoglobulins;
  * Other significant drugs that affect the course of treatment

CONTACTS AND LOCATIONS:
Locations (12):
- Kazakhstan (12):
  - State Enterprise on the Right of Economic Management - Aktobe Medical Center, Aktobe
  - ESEM Pharmacy LLP, Almaty
  - JSC Research Institute of Cardiology and Internal Diseases, Almaty
  - Municipal state enterprise with the right of economic management City polyclinic No. 5, Almaty
  - Non-Profit Joint Stock Company Kazakh National Medical University named after S.D. Asfendiyarov, Almaty
  - Republican Diagnostic Center of Astana Corporate Fund University Medical Center, Astana
  - Municipal State Enterprise on the Right of Economic Management - Pavlodar Regional Hospital named after G. Sultanov, Pavlodar
  - Non-Profit Joint Stock Company Semey Medical University - University Hospital, Semey
  - Medical Center for Joint Diseases of Shymkent LLP, Shymkent
  - State Enterprise on the Right of Economic Management - Regional Clinical Hospital of the Turkestan Region, Shymkent
  - State-owned enterprise on the right of economic management -Taldykorgan City Polyclinic, Taldykorgan
  - Zhambyl Regional Multidisciplinary Hospital of the Health Department of the Akimat of Zhambyl Region, Taraz

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/